CLINICAL TRIAL: NCT04002895
Title: Interventional, Open-label, Single-dose Study Investigating the Absorption, Metabolism and Excretion (AME) of Foliglurax (Lu AF99757) Following Oral Dosing of 14C-foliglurax to Healthy Men
Brief Title: What the Body Does to Foliglurax in Healthy Volunteers
Acronym: Foliglurax
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18154A
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-11-04 (Actual); Status verified 2019-11

CONDITIONS: Healthy
MeSH Terms: interventions — foliglurax

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Foliglurax (Experimental)
  Interventions: Drug: Foliglurax

INTERVENTIONS:
Drug: Foliglurax — Single oral dose of 80 mg [14C]-foliglurax(93µCi/3.44 MBq), 1mg/mL oral solution (prepared from [14C]-foliglurax powder for oral solution)

SUMMARY:
This study evaluates how the body takes up and gets rid of foliglurax after swallowing a liquid dose.

DETAILED DESCRIPTION:
Six healthy men will swallow a liquid dose of 80 mg that is labelled with a small dose of radioactive tracer. Blood, urine and faeces will be collected to measure how much of the radioactivity gets into the blood stream and ends up in the urine and faeces. It is also measured how the body gets rid of the radioactivity and how quickly.

ELIGIBILITY:
Inclusion Criteria:

- Healthy men with a body mass index (BMI) of 19-30 kg/m2 (inclusive), and with a body weight of minimum 60 kg at the Screening Visit.

Exclusion Criteria:

- The subject has or has had any clinically significant immunological, cardiovascular, respiratory, metabolic, renal, hepatic, gastrointestinal, endocrinological, haematological, dermatological, venereal, neurological, or psychiatric disease or other major disorder.

Other inclusion and exclusion criteria may apply.

Ages: 45 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-08 (Actual)

PRIMARY OUTCOMES:
Total amount of radioactivity excreted | Before dosing until day 11
  Cumulative amount of radioactivity excreted in urine and faeces
AUC(0-inf) foliglurax | From day 1 until day 11
  Area under the plasma concentration time curve from zero to infinity
Cmax foliglurax | From day 1 until day 11
  Maximum observed plasma concentration
CL/F foliglurax | From Day 1 until Day 11
  Oral clearance for foliglurax in plasma
Total recovery of the administered dose | Before dosing until day 11
  % of dose in urine and faeces

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@Lundbeck.com
Locations (1):
- GB1050 Covance, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided